CLINICAL TRIAL: NCT01323179
Title: Acute Pain After Fast-track Total Knee Arthroplasty: Preoperative Opioid Versus Non-opioid
Brief Title: Preopioid Versus Nonopioid in Total Knee Arthroplasty (TKA)
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Other Study IDs: 11123111
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Postoperative opioid requirements
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Strong opioids: Patients taking strong opioids preoperatively
- Weak opioids: Patients taking weak opioids preoperatively
- Opioid native: Patients not taking opioids preoperatively

SUMMARY:
Observational study evaluating pain response after total knee arthroplasty (TKA) in patients taking strong, weak or no opioids preoperatively.

ELIGIBILITY:
Inclusion Criteria:

Patients operated with elective, primary, unilateral total knee arthroplasty (TKA) (taking strong or weak opioid daily for minimum 4 weeks or opioid naive patients)

Exclusion Criteria:

* Bilateral / revision arthroplasty
* Disease affection central or peripheral nerve function
* Alcohol and medical abuse
* Daily use of glucocorticoids
* Malignancy
* BMI > 40
* Dementia or other cognitive dysfunction
* Treatment of anxiety or depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated with elective, primary, unilateral total knee artroplasty (TKA).
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours
  Pain during ambulation and at rest

SECONDARY OUTCOMES:
Pain | 7 days
  Pain during ambulation and at rest
Opioid consumption | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Troels H Lunn, MD, Principal Investigator — Dep. of Anesthesiology, Hvidovre University Hospital
Locations (4):
- Denmark (4):
  - Dep. of ortopedic surgery, Gentofte Hospital, Hellerup, Hellerup
  - Dep. of ortopedic surgery, Regionshospitalet Holstebro, Holstebro, Holstebro
  - Dep. of Anesthesiology, Hvidovre University Hospital, Copenhagen, Hvidovre
  - Dep. of ortopedic surgery, Vejle Sygehus, Vejle, Vejle